CLINICAL TRIAL: NCT06162234
Title: Long Term Observation of Ocular Structure and Visual Function in Eyes With High Myopia：Wuhan High Myopia Study
Brief Title: Wuhan High Myopia Study
Acronym: LOVE-WH
Status: Recruiting | Type: Observational
Sponsor: Renmin Hospital of Wuhan University (Other)
Responsible Party: Principal Investigator, Changzheng Chen, Chief of Department of Ophthalmology, Renmin Hospital of Wuhan University
Other Study IDs: WWDRY2023-K074
Record Dates: First submitted 2023-12-01; First posted 2023-12-08 (Actual); Last update posted 2023-12-27 (Actual); Status verified 2023-12

CONDITIONS: High Myopia
Keywords: ocular biometric parameters; Refractive Errors
MeSH Terms: conditions — Refractive Errors | interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Years
Biospecimen Retention: None Retained — tear，saliva
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- entire cohort: entire cohort made up of high myopia patients（observational study）
  Interventions: Other: observational

INTERVENTIONS:
Other: observational — none (observational study)

SUMMARY:
The study aims to observe the long-term changes of ocular（especially fundus） structure and visual function in patients with high myopia, so as to provide evidence for the prevention, diagnosis and prognosis of high myopia.

DETAILED DESCRIPTION:
High myopia is defined as a refractive error of ≤-6.00D or an axial length greater than 26mm. In recent years, the population of highly myopic individuals has been increasing rapidly. Scholars predict that if no effective interventions are taken, the global incidence rate of myopia is expected to increase from 22.9% in 2000 to 49.8% in 2050, and the visual impairment caused by high myopia will be seven times higher than in 2000 on a global scale. In China, a survey conducted by the National Health Commission in 2018 found that highly myopic students accounted for 21.9% of third-year high school students, indicating that high myopia has become a major public health issue due to its prevalence among younger populations.

In recent years, with the development of ocular imaging technologies such as optical coherence tomography (OCT) and corresponding image analysis techniques, high-resolution, non-invasive, fast and in vivo retinal imaging has become more accessible. This has led to the discovery and exploration of various imaging parameters related to optic disc and macula changes in highly myopic patients. We will conduct a 4 years prospective cohort study in the population of 1000 high myopia and controls which have established in mainly college student population, using the latest OCT-A and SS-OCT to observe the long-term changes of fundus structure combined with visual function in patients with high myopia , and explore biomarkers affecting visual function, so as to provide basis for prevention and control of high myopia and prognosis.

ELIGIBILITY:
Inclusion Criteria:

* Voluntarily sign informed consent;
* Commit to follow the research procedures and cooperate with the whole process of the study;
* Age ≥18 years old;
* Best corrected visual acuity ≥0.1;
* Spherical Equivalent Refraction≤-6.00D or axial length ≥26mm in high myopia group；

Exclusion Criteria:

* Unable or unwilling to sign informed consent;
* Unable to cooperate with the examination;
* Astigmatism ≤-1.5D；
* Patients with refractive interstitial opacity so that fundus images cannot be collected；
* Patients with fundus diseases such as diabetic retinopathy, hypertensive retinopathy, age-related macular degeneration, retinal vein obstruction, retinal artery obstruction, etc

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: First-year college student from Wuhan University
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2023-12-25 (Estimated); Primary Completion 2027-09-01 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
Myopic optic nerve changes | Baseline and 6 months and 1，2,3,4years
  Changes in the optic nerve head morphology and blood supply which are supposed to be related with high myopia，examined by fundus photography，OCT，OCTA，etc
Progression of axial length (AL) | Baseline and 6 months and 1，2,3,4years
  Subjects' axial length and its progression collected by IOL master 700
Incidence and progression of visual field (VF) defects | Baseline and 6 months and 1，2,3,4years
  Variety and progression of visual field defects collected by Humphrey 860 perimetry
Loss of best corrected visual acuity（BCVA） | Baseline and 6 months and 1，2,3,4years
  Incidence of BCVA loss collected by subjective optometry
Incidence and progression of myopic maculopathy | Baseline and 6 months and 1，2,3,4years
  Collected by color fundus photography and ultra-wide fundus photography

SECONDARY OUTCOMES:
Relationship between the changes of visual function and pathological changes among patients with high myopia | Baseline and 6 months and 1，2,3,4years
  Relationship between the changes of visual function including best corrected visual acuity and visual field and pathological changes among patients with high myopia
Structural parameters of anterior segment | Baseline and 6 months and 1，2,3,4years
  Structural parameters of anterior segment including corneal curvature，lens thickness(LT)，etc
Intraocular pressure(IOP) | Baseline and 6 months and 1，2,3,4years
  Incidence of elevated intraocular pressure collected by a non-contact tonometer
Mental state and quality of life | Baseline and 6 months and 1，2,3,4years
  Mental state and quality of life collected by a questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Renmin Hospital of Wuhan University, Wuhan, Hubei, China